CLINICAL TRIAL: NCT07402681
Title: Evaluating Symptom Variations and Observing Longitudinal Individual Change Effects in TF-CBT
Acronym: EVOLVE
Status: Recruiting | Type: Observational
Sponsor: University Children's Hospital, Zurich (Other)
Collaborators: Otto-Friedrich-University Bamberg (Other); Catholic University of Eichstätt-Ingolstadt (Other)
Responsible Party: Principal Investigator, Lasse Bartels, Postdoctoral fellow, University Children's Hospital, Zurich
Other Study IDs: 2024-00903
Record Dates: First submitted 2026-01-13; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Post-traumatic Stress Symptoms
Keywords: TF-CBT; post-traumatic stress symptoms; single-case experimental design

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Trauma-focused Cognitive Behavioral Therapy for Children and Adolescents — TF-CBT is a child and family-focused, component-based trauma-focused intervention that aims to address post-traumatic stress symptoms and other trauma-related difficulties (e.g., anxiety, depression) associated with traumatic events.

SUMMARY:
The goal of this observational study is to learn about the level of change in post-traumatic stress symptoms in adolescents with traumatic experiences over the course of trauma-focused cognitive behavioral therapy for children and adolescents according to Cohen, Manarinno, & Deblinger (2017).

ELIGIBILITY:
Participants will be included if:

1. they are between 12 and 18 years of age;
2. they have been exposed to at least one or more traumatic event(s) according to the DSM-5 A criteria after the age of 3 years and dating back at least 1 months (with regard to the ability of patients to remember the event(s) and to the high spontaneous remissions of PTSS in the first month after a traumatic event);
3. they exhibit high severity of DSM-5 PTSS as indicated by a total symptom score of ≥25 assessed with the Child and Adolescent Trauma Screen 2 (CATS-2);
4. a nonoffending adult caregiver is available for the treatment and willing to participate in weekly treatment sessions (the inclusion of a caregiver is integral to the TF-CBT treatment model);
5. they are willing and able to attend weekly treatment sessions;
6. if their living circumstances are safe and stable to minimize the risk of re-traumatization during the project;
7. they and their caregiver have sufficient command of the German language (i.e., to participate in assessment [read] and treatment[converse]);
8. they and their caregivers possess a smartphone.
9. they and their caregiver provided written informed consent.

Participants will not be included if:

1. they exhibit acute suicidal behavior or have suicidal ideations requiring immediate hospitalization;
2. they have a documented developmental disorder (i.e., autism spectrum disorder) or current psychosis based on adolescent- and caregiver-report and clinical assessment;
3. they exhibit severe substance misuse based on clinical assessment;
4. take part in concurrent psychotherapy during TF-CBT;
5. exhibit severe intellectual disability based on clinical assessment.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents between 12 and 18 years for whom trauma-focused treatment is indicated due to a PTE/ PTEs they have experienced as well as a significant level of PTSS.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Short, semi-individually-tailored questionnaire - so-called Idiosyncratic Assessment (IA) - assessing the six ICD-11 PTSS plus six individually selected PTSS that are most distressing to the patient. | The IA will be assessed every two days four weeks before the start of TF-CBT treatment as well as every two days over the course of TF-CBT treatment; up to 1year
  The 12 symptoms are selected at the baseline assessment from the Child And Adolescent Trauma Screen 2 (Sachser et al., 2022). A Visual Analogue Scale is utilized the intensity of symptoms (0 = not at all - 100 = extreme)

SECONDARY OUTCOMES:
International Depression Questionnaire (IDQ) | Baseline, pre-treatment, after TF-CBT stabilization and skills phase, after TF-CBT trauma narrative treatment phase, after TF-CBT cognitive restructuring-treatment phase, post-treatment, three-month follow-up; up to 1.5 years
  ICD-11 single episode depressive disorder (self- and Caregiver-report); score range: 0 - 27; higher scores mean worse outcome.
International Anxiety Questionnaire (IAQ) | Baseline, pre-treatment, after TF-CBT stabilization and skills phase, after TF-CBT trauma narrative treatment phase, after TF-CBT cognitive restructuring-treatment phase, post-treatment, three-month follow-up; up to 1.5 years
  ICD-11 generalised anxiety disorder (self- and caregiver-report); score range: 0 - 24; higher scores mean worse outcome.
Child Post-Traumatic Cognitions Inventory (CPTCI) | Baseline, pre-treatment, after TF-CBT stabilization and skills phase, after TF-CBT trauma narrative treatment phase, after TF-CBT cognitive restructuring-treatment phase, post-treatment, three-month follow-up, up to 1.5 years
  Negative trauma-related cognitions (self-report); ranges are from 25 to 100 for the total scale; higher scores indicate more dysfunctional trauma-related cognitions.
Child and Adolescent Trauma Screen 2 (CATS-2) | Baseline, pre-treatment, after TF-CBT stabilization and skills phase, after TF-CBT trauma narrative treatment phase, after TF-CBT cognitive restructuring-treatment phase, post-treatment, three-month follow-up, up to 1.5 years
  Potentially traumatic events; DSM-5/ICD-11 post-traumatic stress symptoms (self- and caregiver-report); total score range: 0-60; higher scores mean worse outcome.
Functioning scale of the Ohio Scales Youth Scales | Baseline, pre-treatment, after TF-CBT stabilization and skills phase, after TF-CBT trauma narrative treatment phase, after TF-CBT cognitive restructuring-treatment phase, post-treatment, three-month follow-up, up to 1.5 years
  Level of daily functioning (self- and caregiver-report); score range: 0-80 higher scores mean better outcome.
Inventory for the assessment of Negative Effects of Psychotherapy for children and adolescents | Post-treatment, up to 1 year
  Unwanted negative effects of psychotherapy (self- and caregiver-report); score range: 0-54; higher scores mean worse outcome.
Parental Acceptance Rejection Questionnaire (PARQ) | Baseline, pre-treatment, after TF-CBT stabilization and skills phase, after TF-CBT trauma narrative treatment phase, after TF-CBT cognitive restructuring-treatment phase, post-treatment, three-month follow-up, up to 1.5 years
  Interpersonal acceptance and rejection in the child-parent relationship (self- and caregiver-report); score range: 24-96; higher scores mean worse outcome.
Session Rating Scale (SRS) | After every TF-CBT treatment session, up to 1 year
  Therapeutic Relationship (self-report); score range: 0-40; higher scores mean better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- University Children's Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided